CLINICAL TRIAL: NCT03976596
Title: Measurement of in Vivo Mitochondrial Capacity in Infants: a 31P-MRS Pilot Study
Brief Title: Measurement of in Vivo Mitochondrial Capacity in Infants
Status: Terminated | Type: Observational
Why Stopped: Decoupler equipment used for 31P magnetic resonance is being serviced
Sponsor: Pennington Biomedical Research Center (Other)
Responsible Party: Principal Investigator, Leanne Redman, Associate Professor, Pennington Biomedical Research Center
Other Study IDs: PBRC 2018-051
Record Dates: First submitted 2019-06-04; First posted 2019-06-06 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-02

CONDITIONS: Healthy Infants
Keywords: neonates; mitochondria; MRI

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The overarching aim of this project is to determine the test re-test reliability of 31P-magnetic resonance spectroscopy measurements in infants. Primary endpoints include two separate measures of in vivo mitochondrial capacity (ATPmax) over a 1-10 day period to assess feasibility and reliability.

ELIGIBILITY:
Inclusion Criteria:

* healthy, full-term infant
* aged 14-28 days at Visit 1
* willingness of parents to be notified of incidental findings from study procedures

Exclusion Criteria:

* born preterm
* implanted metal or electronic objects that render MRI unsafe
* unable to complete 2 clinic visits 1-10 days apart at Pennington Biomedical Research Center

Ages: 14 Days to 28 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: This cross-sectional study will enroll up to 18 infants. Infants will complete 2 study visits over a 1-10 day period for outcome measures.
Sampling Method: Non-Probability Sample
Enrollment: 2 (Actual)
Dates: Start 2019-05-21 (Actual); Primary Completion 2019-07-02 (Actual); Study Completion 2019-07-02 (Actual)

PRIMARY OUTCOMES:
In vivo mitochondrial capacity (ATPmax) | 1 day
  In vivo mitochondrial capacity as measured by phosphorus magnetic resonance spectroscopy

CONTACTS AND LOCATIONS:
Overall Officials: Leanne M Redman, PhD, Principal Investigator — Pennington Biomedical Research Center
Locations (1):
- Pennington Biomedical Research Center, Baton Rouge, Louisiana, United States

IPD SHARING:
Plan to Share IPD: No